CLINICAL TRIAL: NCT00207038
Title: Airway Inflammation in Swimmers: Development and Risk Factors
Brief Title: Airway Inflammation in Swimmers
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Imperial College London (Other); Sygekassernes Helsefond (Other); Toyota-Fonden (Other); Team Denmark (Other); Anti Doping Danmark (Other); Ragnhild Ibsens Legat For Medicinsk Forskning (Other); Kong Christian IX og Dronning Louises Jubilæumslegat (Unknown); Kong Christian den Tiendes Fond (Unknown)
Responsible Party: Lars Pedersen, Bispebjerg Hospital
Other Study IDs: (KF) 01 261528
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Asthma
Keywords: Asthma; Airway inflammation; Sport
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples EBC Sputum

SUMMARY:
Studies have shown that the prevalence of respiratory symptoms, airway hyperresponsiveness (AHR) and asthma is high and increasing in elite athletes. The inflammation seen in the airways of elite athletes might differ from the inflammation seen in the airways of "ordinary" asthmatics and it might represent a different kind of asthma.

The primary purposes are

1. To investigate the type of airway inflammation in young swimmers.
2. To investigate the acute changes in airway inflammation after a short training session.

ELIGIBILITY:
Inclusion Criteria:

* Swimmer

Exclusion Criteria:

* Current smoker or more than 3 pack-years

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Elite swimmers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2005-09; Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Pedersen, MD, Study Chair — Respiratory and Allergy Reseach Unit, Department of Internal Medicine, Bispebjerg Bakke 23, Bispebjerg Hospital, University Hospital of Copenhagen, DK-2400 Copenhagen NV, Denmark
Locations (1):
- Respiratory and Allergy Research Unit, Department of Internal Medicine, Bispebjerg Hospital, University Hospital of Copenhagen, Copenhagen, Denmark